CLINICAL TRIAL: NCT00709202
Title: The Attenuation of Second Generation Antipsychotic Induced Weight Gain in Adolescents and Adults Using Betahistine: A Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy and Tolerability Study of Betahistine to Ameliorate Antipsychotic Associated Weight Gain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Robert C. Smith MD PhD, Research Psychiatrist, Research Professor of Psychiatry, Nathan Kline Institute for Psychiatric Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07TGF-1112
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Bipolar I Disorder; Bipolar II; Bipolar NOS(Not Otherwise Specified); Psychotic Disorder Not Otherwise Specified; Autism Spectrum Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Autism Spectrum Disorder | interventions — Betahistine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subjects assigned to this arm will receive Betahistine.
  Interventions: Drug: Betahistine
- 2 (Placebo Comparator): Subjects in this group will received placebo.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Betahistine — Subjects will be started on 8 mg BID of Betahistine and titrated up to 24 mg BID (BID = 2 times a day)..
  Other Names: Serc, Betaserc, Betaserk
  Arms: 1
Drug: Placebo Oral Tablet
  Arms: 2

SUMMARY:
The study attempts to evaluate a histamine analog long used for the treatment of Meniere's disease, betahistine, that shows promise in reversing the antihistaminergic effects thought to be involved in antipsychotic induced weight gain.

Hypothesis to be tested:

A. Patients who have gained a developmentally inappropriate amount of weight on antipsychotics (AP) will see their weight and BMI decrease with betahistine augmentation as compared to placebo augmentation.

B. Betahistine augmentation in AP treated patients will increase levels of satiety in a standardized meal situation and decrease caloric intake as compared to placebo augmentation.

C. Metabolic effects of betahistine augmentation in AP treated patients will be reflected in differences in waist circumference, hip circumference and waist hip ratios D. Betahistine augmentation in this population will lead to decrease in fasting glucose-lipid lab values related to the development of metabolic syndrome as compared to placebo augmentation

DETAILED DESCRIPTION:
Subjects for this study were adolescents and adults from age 12 to age 59. Subjects were individuals who have been psychiatrically stabilized on first or second generation antipsychotic medication, and have gained substantial weight during their treatment. Subjects were excluded if they have asthma, peptic ulcer disease (diseases which may be exacerbated by a histamine analog) or are prescribed medications known to affect body composition or metabolism other than those currently being studied. Subjects were randomized to receive either betahistine or placebo at a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and Adults ages 12-59 with a diagnosis of Schizophrenia, Schizoaffective Disorder, Schizophreniform, Bipolar I, Bipolar II, Bipolar NOS or Psychotic Disorder NOS, Autism Spectrum Disorder
* Patients will be currently treated with antipsychotics

Patients will qualify for entry if they meet the following weight criteria:

1. The patient has gained 7% of their weight since beginning of treatment with one or more of the current antipsychotics.
2. The patient has had an increase of 7% of their weight during the last year while being treated with antipsychotics.
3. The patient has a BMI of 30 or more and has gained 10 lbs or more in the past 8 months while being treated with antipsychotic medications.
4. The patient has a BMI of 35 or greater at the current time, and his chart shows a history of consistent weight gain over the past 1 to 3 years during treatment with antipsychotics.

   .

   Exclusion Criteria:
   * Subjects will be excluded if they have asthma, peptic ulcer disease (diseases which may be exacerbated by a histamine analog), or history of pheochromocytoma or peptic ulcer disease. Patients will be excluded if they are prescribed medications known to affect body weight or glucose-lipid metabolism, such as prescription or over the counter medications taken for the purpose of weight reduction. Subjects who are currently treated with metformin, for less than 6 months and have shown recent weight change on metformin. Patients on thyroid replacement therapy or lipid-lowering agents whose dosage has changed by more than 50 % in the past month will be excluded. If they are relatively stable doses of these medications they will not be excluded. Patients who are on lipid lowering medication, thyroid replacement medication, or diabetes medication, (excluding metformin), must remain on these medications throughout the period of the study. Females who are pregnant or breast feeding will be excluded.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-07; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Smith, M.D., Principal Investigator — Nathan Kline Institute for Psychiatric Research
Locations (1):
- Nathan Kline Insitute for Psychiatric Research, Orangeburg, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang D, Jing Z, Li R, Hei G, Shao T, Li L, Sun M, Yang Y, Wang Y, Wang X, Long Y, Huang X, Wu R. Effect of Betahistine and Metformin on Antipsychotic-Induced Weight Gain: An Analysis of Two Clinical Trials. Front Psychiatry. 2018 Nov 27;9:620. doi: 10.3389/fpsyt.2018.00620. eCollection 2018. PMID 30542300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 48 subjects signed consent for the study. 8 subjects withdrew consent before randomization and another subject withdrew before the first post-baseline measurement. Therefore, only 39 subjects were analyzed.
Groups:
- Betahistine: Subjects assigned to this arm will receive Betahistine.
  Betahistine: Subjects will be started on 8 mg BID of Betahistine and titrated up to 24 mg BID.
- Placebo: Subjects in this group will received placebo.
  Placebo: Subjects will be receive placebo tablets matched in number to betahistine tablets
Period: Overall Study
Arm/Group | Betahistine | Placebo
Started | 19 | 21
Completed | 13 | 15
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 6 | 6

BASELINE CHARACTERISTICS:
Population: One subject randomized to placebo group discontinued participation before the first post-baseline measurement, and, therefore, eh was not considered as relevant in the analysis of data. Therefore, background data is presented on 39 of the 40 subjects who were analyzed for outcome variables.
Groups:
- Placebo: Subjects in this group will received placebo.
  Betahistine: Subjects will be started on 8 mg BID of Betahistine and titrated up to 24 mg BID.
- Total: Total of all reporting groups
Arm/Group | Betahistine | Placebo | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data is presented on 39 subjects who had data sufficient data for analysis of variables of clinical interest-who received at least one post baseline evaluation. One subject discontinued shortly after randomization assignment.
  years | 31.1 (14.9) | 31.1 (14.0) | 31.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 7 | 9 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race-Ethnicity based on Self-Description of participants. Other category involves participants with middle eastern or other background who could not give precise ethnic description.
  Participants
    Race-Ethnicity: White-Caucasian | 4 | 9 | 13
    Race-Ethnicity: Black-African American | 7 | 7 | 14
    Race-Ethnicity: Hispanic | 4 | 4 | 8
    Race-Ethnicity: Other | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Least Squares estimated change in weight from end of study minus baseline
Time Frame: Measured at each visit from baseline to end of study over a 12 week period
Population: Least Squares estimated change in weight from end of study minus baseline for all subjects who had at least one post-baseline weight evaluation, using mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: kg. (killograms)
Groups:
- Placebo: Subjects in this group will received placebo.
  Placebo Oral Tablet
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 19 | 20
kg. (killograms) | -2.0021 (0.7970) | -1.5490 (0.7650)

2. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Least Squares estimated change in BMI from end of study minus baseline
Time Frame: Measured at each visit from baseline to end of study over a 12 week period.
Population: Least Squares estimated change in BMI from end of study minus baseline for all subjects who had at least one post-baseline weight evaluation, using mixed model analysis.
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 19 | 20
kg/m^2 | -0.5524 (0.2747) | -0.5637 (0.2653)

3. Secondary Outcome: Change in Waist Circumference
Description: Least Squares estimated change in waist circumference from end of study minus baseline
Time Frame: Measured at each visit from baseline to end of study over a 12 week period.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 19 | 20
centimeters | 4.0928 (1.3884) | 2.4864 (1.3669)

4. Secondary Outcome: Change in Hip Circumference
Description: Least Squares estimated change in hip circumference from end of study minus baseline
Time Frame: Measured at each visit from baseline to end of study over a 12 week period.
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 19 | 20
centimeters | 1.7957 (1.3837) | 1.3668 (1.3118)

5. Secondary Outcome: Change in Glucose
Description: Least Squares estimated change in glucose from end of study minus baseline
Time Frame: Measured at each visit from baseline to end of study over a 12 week period.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 14 | 14
mg/dL | 4.292 (2.116) | 3.136 (2.116)

6. Secondary Outcome: Change in Cholesterol
Description: Least Squares estimated change in cholesterol from end of study minus baseline
Time Frame: Measured at each visit from baseline to end of study over a 12 week period.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 14 | 14
mg/dL | 1.087 (0.079) | 1.010 (0.079)

7. Secondary Outcome: Change in LDL
Description: Least Squares estimated change in LDL from end of study minus baseline
Time Frame: Measured at each visit from baseline to end of study over a 12 week period.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 14 | 14
mg/dL | 1.799 (6.633) | 0.915 (6.633)

8. Secondary Outcome: Change in HDL
Description: Least Squares estimated change in HDL from end of study minus baseline
Time Frame: Measured at each visit from baseline to end of study over a 12 week period.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 14 | 14
mg/dL | 2.555 (1.815) | -0.840 (1.815)

9. Secondary Outcome: Change in Triglycerides
Description: Least Squares estimated change in triglycerides from end of study minus baseline
Time Frame: Measured at each visit from baseline to end of study over a 12 week period.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 14 | 14
mg/dL | -4.426 (11.119) | -3.360 (11.119)

10. Secondary Outcome: Change in Appetite Hunger
Description: Least Squares estimated change in appetite hunger from end of study minus baseline.The scale used has no specific name. It is a Visual Analogue Scale, where a line is drawn of 10 cm long with the statement beneath the line" How Hungry do you feel '. The subject places an X on the line. The measurements, the number of centimeters from the start of the line ("O"), indicate the amount of hunger. The higher the cm number the higher the feeling of hunger. The measure reported is the difference in this scale reading in cm from after the test meal to before consuming the test meal. The number (mean, s.e.m) presented is the analysis of covariance model estimated difference score at the end of study, with the covariate of the same score at baseline.
Time Frame: Measured at baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 14 | 17
units on a scale | -3.605 (.896) | -3.684 (.813)

11. Secondary Outcome: Change in Appetite Fullness
Description: Least Squares estimated change in appetite fullness from end of study minus baseline.The scale used has no specific name. It is a Visual Analogue Scale, where a line is drawn of 10 cm long with the statement beneath the line" How full do you feel '. The subject places an X on the line. The measurements, the number of centimeters from the start of the line ("O"). indicate amount of feeling of fullness. The higher the cm number the higher the feeling of fullness. The measure reported is the difference in this scale reading in cm from after the test meal to before consuming the test meal. The number (mean, s.e.m.) presented is the analysis of covariance model estimated difference score at the end of study, with the covariate of the same score at baseline.
Time Frame: .Measured at baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Betahistine | Placebo
Number analyzed (Participants) | 13 | 17
units on a scale | 1.800 (1.058) | 4.698 (.925)

ADVERSE EVENTS:
Time Frame: 12 weeks during study drug administration
Description: We are reporting adverse events reported to IRB (Institutional Review Board) on adverse event forms.
Arm/Group | Betahistine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 2/19 | 4/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Betahistine (N=19) | Placebo (N=20)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Vomited after session which included drinking vanilla milkshake. No sequelae.
conjunctivitis (Eye disorders) | 1 (1) | 0 (0) — Conjunctivitis (Pink Eye) developed in week 2 of study. Successfully treated with Ciprofloxacin
chest pain (Cardiac disorders) | 0 (0) | 1 (1) — Chest pain and shortness of breath. Medical examination and labs for pulmonary embolism and cardiac enzymes levels were normal..
skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Exfoliated skin rash over sun exposed neck area.
chest pain (Psychiatric disorders) | 0 (0) | 1 (1) — Patient was psychiatrically evaluated for what mother described as difficult behavior after sexual assault.
Increase in level of psychiatric symptoms (Psychiatric disorders) | 0 (0) | 1 (1) — Patient had increase in level of hallucinations, unusual thought content, and suspicious on Brief Psychiatric Rating Scale.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No